CLINICAL TRIAL: NCT04628897
Title: Risk Factors for Low Physical Activity Levels in Preschool-aged Children in a Densely Populated Urban Community in Bangladesh
Brief Title: Physical Activity and the Home Environment in Preschool-aged Children in Urban Bangladesh
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Roth, Principal Investigator, The Hospital for Sick Children
Other Study IDs: 1000057061
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Obesity, Childhood; Malnutrition; Anemia
Keywords: Obesity; Home Environment; Malnutrition
MeSH Terms: conditions — Pediatric Obesity; Malnutrition; Anemia; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Exposures — 1. Total area of available floor space inside the home (m2)
  2. Frequency that child plays outdoors
  3. Total number of physical hazards in the home (presence of open stairwells, stove height)
  4. Total number of fine-motor activity items available to the child
  5. Presence of gross-motor activity items available to the child across each category (e.g., fixed, portable: ball equipment, push/pull equipment, riding equipment, rocking and twisting equipment)
  6. Hemoglobin concentration (g/L).

SUMMARY:
The overall goal of this study is to generate new knowledge regarding the nutritional and environmental determinants of physical activity in young children living in a densely populated urban community in Bangladesh. The investigators hypothesize that low levels of preschooler physical activity are associated with a lack of play-oriented physical attributes (i.e., total area of indoor floor space, presence and count of unsafe physical hazards, and presence and count of stationary and portable gross motor activity-oriented items) within the homes in urban Bangladesh. The investigators also hypothesized that low Hb may be associated with low physical activity levels in this population.

DETAILED DESCRIPTION:
Study Rationale

As the double burden of nutrition emerges in Bangladesh and other low- to middle-income countries, it is imperative to develop strategies to mitigate the adverse effects associated with both undernutrition and obesity. Identifying levels of physical activity among children is a requisite step to developing and targeting interventions to promote physical activity among young populations. Furthermore, exploring the risk factors associated with physical activity levels in young children can help better inform policy makers surrounding a public health intervention.

Goals The overall goal of the research is to generate new knowledge regarding the nutritional and environmental determinants of physical activity in young children living in a densely populated urban community in Bangladesh.

Primary Objectives

The specific objectives of this study are to:

1. Describe physical activity levels in a sample of preschool-aged children in an inner-city community in Dhaka, Bangladesh,
2. Estimate the associations between characteristics of the physical environment of the home (total area of available floor space inside of the home, number and presence of physical hazards, and the number of gross motor activity-oriented items present) and the physical activity levels of preschoolers in Dhaka, and
3. Estimate the associations between hemoglobin concentration (Hb) and preschooler physical activity level.
4. Describe sleep quantity and quality in the sample of preschool-aged children in urban Bangladesh

The investigators conducted a cross-sectional observational study of preschool-aged children between 34-38 months of age (n=60) selected from the ongoing Maternal Vitamin D for Infant Growth (MDIG) trial cohort (NCT01924013) in Dhaka, Bangladesh. The investigators planned to enrol a minimum of 60 participants with complete data sets, with recruitment up to 90 participants until this enrolment target was reached.

Study Procedures

* Accelerometry
* Home built environment audit
* Anthropometry
* hemoglobin concentration
* Maternal perception of the home environment and household food security

ELIGIBILITY:
Inclusion Criteria:

* Child is 34-38 months of age;
* Child and primary caregiver reside in Dhaka or urban environs;
* Parent/guardian provides written informed consent for study procedures.

Exclusion Criteria:

* Child requires mobility assistance and/or has been diagnosed with a major neurological or orthopedic condition or disorder affecting physical activity (e.g., cerebral palsy, club foot, etc.).
* Major physician-diagnosed chronic respiratory or cardiac disease that limits physical activity (e.g., severe asthma, currently taking medication for symptomatic congenital heart disease, etc.).

Ages: 34 Months to 38 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants within the Maternal Vitamin D for Infant Growth (MDIG) trial (NCT01924013) cohort registry who have a) expressed interest in participating in future sub-studies, and b) have children within the target age range, will be contacted. Participants will be contacted prior to their anticipated study visit. A contact list will be updated each week to prospectively recruit participants in advance or during the age window in which children are eligible for enrolment. Each list will begin with the eldest children to reduce the number of missed opportunities to enroll children before they exit the eligible age window. The catchment area will include the following neighbourhoods in urban Dhaka: Kamrangir char, Azimpur, Lalbag, and Hazariba
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-09-17 (Actual); Primary Completion 2017-12-09 (Actual); Study Completion 2017-12-09 (Actual)

PRIMARY OUTCOMES:
Moderate-to-Vigorous Physical Activity | 3-14 days
  Objectively measured accelerometry data, a continuous variable reflecting mean daily PA during the study period, expressed as mean counts per 15 seconds (cp15s). This summary measure was generated by first calculating mean daily PA, then averaging the daily means across collection days, including data between the time the child woke up until the time the child went to sleep, as reported by the caregiver on all days that met criteria for inclusion (i.e., at least 10 hours of wear time)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roth, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Details of the data sharing plan are still to be determined.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: To be determined
Access Criteria: To be determined

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT04628897/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT04628897/ICF_001.pdf